CLINICAL TRIAL: NCT00985205
Title: Effects of Enteral Glutamine Supplementation on Mortality and Infectious Morbidity in Severely Burned Patients: a Multi-center Pilot Trial
Brief Title: The RE-ENERGIZE Study: RandomizEd Trial of ENtERal Glutamine to minimIZE Thermal Injury
Acronym: RE-ENERGIZE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Daren K. Heyland (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Daren K. Heyland, Professor of Medicine, Clinical Evaluation Research Unit at Kingston General Hospital
Organization: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RE-ENERGIZE; CIHR # 190808 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2009-09-25; First posted 2009-09-28 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Burns
Keywords: Randomized Clinical Trial; Glutamine; Themal Burn Injuries; Nutrition; Outcome Assessment; Critical Care; Total Body Surface Area
MeSH Terms: conditions — Burns | interventions — Glutamine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enteral Glutamine (Experimental): 0.5 g/kg/day mixed in water and given via nasogastric or feeding tube as boluses q 4 hrs or TID or QID if po
  Interventions: Dietary Supplement: Enteral Glutamine
- Placebo (Placebo Comparator): Mixed in with water and given via nasogastric or feeding tube as boluses q 4hrs or TID or QID if po
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Enteral Glutamine — 0.5g/kg/day powdered glutamine to be mixed in with water and given via nasogastric or feeding tube q4 hrs or TID or QID if po.
  Other Names: Glutamine
  Arms: Enteral Glutamine
Dietary Supplement: Placebo — Maltodextrin mixed with water given via NG or feeding tube Q 4 hours or TID or QID if po.
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
The purpose of this study is to test the following hypotheses:

1. Enteral glutamine administration decreases in-hospital mortality in adult patients with severe thermal burn injuries.
2. Enteral glutamine administration decreases hospital-acquired blood stream infections from Gram negative organisms and length of stay in ICU and hospital for adult patients with severe thermal burn injuries.
3. Enteral glutamine administration will improve the physical function of surviving burn injured patients and reduce their cost of care.

The objectives of this trial are to determine the overall treatment effect and safety of glutamine in burn patients. Specifically, the investigators want to assess the following outcomes in a sample of 1200 patients in 80 sites:

1. In patients with severe, life-threatening burn injury, what is the effect of enteral glutamine on time to discharge alive from hospital
2. In patients with severe, life-threatening burn injury, what is the effect of enteral glutamine on 6 month mortality, hospital-acquired blood stream infections from Gram negative organisms, hospital mortality, duration of stay in ICU and hospital, health-related quality of life, and health care resources?

DETAILED DESCRIPTION:
Burn injuries represent a public health problem worldwide, ranked fourth in all injuries and are among the leading cause of disability adjusted life years in low and middle-income countries. More than in any other injury, the inflammation and catabolism associated with severe burns can exacerbate nutrient deficiencies, thereby predisposing patients to impaired immune function and increased risk of developing infectious complications, organ dysfunction, and death. Consequently, over the last few decades numerous trials have evaluated the impact of different nutrition/nutrient strategies in severe burns patients. Glutamine is of particular interest in this regard as it appears vital for a number of key stress-response pathways in serious illness. The existing randomized trials of glutamine supplementation in burns patients have suggested a significant reduction in mortality, infection, and hospital length of stay. However, in other critically ill patient populations, there is a signal of increased mortality associated with glutamine administration. Given this conflicting evidence, burn practitioners are either harming or saving lives with glutamine use. We hypothesize that the inexpensive therapeutic strategy tested in this multicenter randomized controlled clinical trial of supplemental enteral glutamine in 1200 severe burn injury patients will lead to lower morbidity and mortality and reduced health care costs in an otherwise very devastating and disabling injury worldwide.

In our pilot study (Critical Care Medicine, 2003, 31:2444) we found a protective effect of glutamine against blood infection in severely burned adult patients. In addition, a significant decrease in mortality was observed with glutamine. These results should be tested with a multi-center trial because our study was small and did not have mortality as an end point.

The specific aims of the study are to determine the overall treatment effect and safety of glutamine in burn patients. Clinical outcomes will be: mortality, time to discharge alive, incidence of acquired bacteremia due to Gram negative organisms, hospital mortality, duration of mechanical ventilation, ICU stay and hospital stay. The cost-effectiveness of glutamine administration will also be measured if the results show a decrease in length of care or a reduced incidence of acquired bacteremia due to Gram negative organisms with glutamine.

The study will be a large, multicenter, double-blind, pragmatic, randomized controlled trial of 1200 patients with severe burns randomly allocated to receive enteral glutamine or placebo. Randomization will be concealed and stratified by site allocating patients 1:1 to either glutamine or matching placebo by the method of permuted blocks of random undisclosed size within strata. Patients will be adults, a minimum of 18 years old, with deep 2nd and/or 3rd degree burns requiring grafting, and for patients age 18 - 39 years a (Total Body Surface Area) TBSA burn ≥ 20% or in the presence of an inhalation injury a minimum of 15% TBSA burn is required; for patients age 40 - 59 years a TBSA burn ≥ 15% is required; for patients aged 60 years or older a TBSA burn ≥ 10% is required. The study will include approximately 80 burn centers in Canada, the US, Europe and Latin America. Patients will receive glutamine or a placebo through their feeding tube, every 4 hours or TID or QID if taking things by mouth, for a total of 0.5 g/kg/day for patients with a BMI <35. Patients with a BMI ≥35 will receive 0.5 g/kg/day based on an obesity-adjusted body weight. The study intervention will be administered until ≥7 days after the last successful grafting operation or until discharge from acute care unit or 3 months from admission, whichever comes first. Resuscitation, nutritional support, pain management, infection control and surgical care will be done according to standardized procedures.

The Data will be collected and managed by a professional and centralized organization for multi centres clinical research (Clinical Evaluation Research Unit, Kingston, Ontario, Canada).

ELIGIBILITY:
Inclusion Criteria:

1. Deep 2nd and/or 3rd degree burns requiring grafting
2. Patient meets one of the following 4 criteria:

   1. Patients 18 - 39 years of age with ≥ 20% TBSA* burn
   2. Patients 18 - 39 years of age with ≥ 15% TBSA* burn and with inhalation injury
   3. Patients 40 - 59 years of age with ≥ 15% TBSA* burn
   4. Patients ≥ 60 years of age ≥ 10% TBSA* *TBSA - Total Body Surface Area

Exclusion Criteria:

1. > 72 hrs from admission to ICU to time of consent.
2. Patients younger than 18 years of age.
3. a) Patients without known renal disease and renal dysfunction defined as a serum creatinine >171 µmol/L or a urine output of less than 500 mL/last 24 hours (or 80 mL/last 4 hours if a 24 hour period of observation is not available).

   b) Patients with acute on chronic renal failure (pre-dialysis) with an absolute increase of >80 µmol/L from baseline or pre-admission creatinine or a urine output of <500 mL/last 24 hours (or 80 mL/last 4 hours).

   c) Patients with chronic renal failure on dialysis will be excluded.
4. Liver cirrhosis - Child-Pugh class C liver disease
5. Pregnant or lactating females.
6. Contra-indication for EN: intestinal occlusion or perforation, intra-abdominal injury.
7. Patients with injuries from high voltage electrical contact.
8. Patients who are moribund (not expected to survive the next 72 hours).
9. Patients with extreme body sizes: BMI < 18 or > 50
10. Enrollment in another industry sponsored ICU intervention study.
11. Received glutamine supplement for > 24 hrs prior to randomization
12. Known allergy to maltodextrin, corn starch, corn, corn products or glutamine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1201 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Time to Discharge Alive | 3 months

SECONDARY OUTCOMES:
6 Month Mortality | 6 Months

OTHER OUTCOMES:
Health-Related Quality of Life - in particular the physical function domain of the SF-36, ADL, and IADL questionnaires. | 6 Month
Incidence of acquired bacteremia due to Gram negative organisms | 3 Months
Hospital Mortality | 3 Months
Duration of Mechanical Ventilation | 3 months
ICU Stay | 3 Months
Hospital Stay | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Daren Heyland, MD, Principal Investigator — Queen's University
Locations (53):
- United States (27):
  - University of South Alabama Medical Center, Mobile, Alabama
  - Arizona Burn Center at Maricopa Medical Center, Phoenix, Arizona
  - Southern California Regional Burn Ctr at LAC & USC Med. Ctr., Los Angeles, California
  - Shriners Hospitals for Children Northern California, Sacramento, California
  - Department of Anesthesiology, University of Colorado, Aurora, Colorado
  - North Colorado Medical Center - Banner Health, Greeley, Colorado
  - Connecticut Burn Center, Bridgeport, Connecticut
  - The Burn Center at Washington Hospital Center, Washington D.C., District of Columbia
  - Shands Burn Center at the University of Florida, Gainesville, Florida
  - University of South Florida/Tampa Gen. Hosp. Reg. Burn Center, FL, Tampa, Florida
  - Joseph M Still Burn Center, Augusta, Georgia
  - Department of Surgery University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Mercy Hospital St. Louis, St Louis, Missouri
  - CHI St.Elizabeth Regional Burn Center, Lincoln, Nebraska
  - The Nebraska Medical Center, Omaha, Nebraska
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Akron's Children's Hospital, Paul & Carol David Foundation, Akron, Ohio
  - The Ohio State University Wexnar Medical Center, Columbus, Ohio
  - Legacy Emmanuel Hospital & Health Center, Portland, Oregon
  - The Western Pennsylvania Hospital Burn Center, Pittsburgh, Pennsylvania
  - Firefighters' Regional Burn Center TN, University of Tennesse Health & Sciences Center, Memphis, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - JBSA Fort Sam Houston, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann/UTHSC, Houston, Texas
  - Harbourview Medical Center, Seattle, Washington
  - Columbia-St. Mary's, Milwaukee, Wi, Milwaukee, Wisconsin
- Medical University of Graz, Graz, Styria, Austria
- Belgium (2):
  - Ghent University Hospital, Ghent
  - University Hospital of Liège, Liège
- The Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil
- Canada (5):
  - Foothills Medical Centre, Calgary, Alberta
  - HHS/Hamilton Firefighters Burn Unit, Hamilton, Ontario
  - Ross Tilley Burn Centre, Sunnybrook Health Sciences Centre, Toronto, Ontario
  - CHUM/Centre des Grands Brules, Montreal, Quebec
  - HEJ/Centre des Grands Brules, Québec
- Instituto Tecnologico de Santo Domingo, Santo Domingo, Dominican Republic
- Germany (2):
  - RWTH Aachen University, Aachen, North Rhine-Westphalia
  - Berufsgenossenschaftliche Unfallklinik Ludwigshafen, Ludwigshafen, Rhein
- A.O.U. Citta della Salute e della Scienza di Torino, Torino, TO, Italy
- Centro Nacional de Quemaduras y Cirugia Reconstructiva, Asunción, Paraguay
- Singapore General Hospital, Singapore, Singapore
- Hospital Universitario La Fe, Valencia, Spain
- Uppsala University Hospital, Uppsala, Sweden
- Thailand (3):
  - Siriraj Hospital, Divison of Trauma Surgery, Mahidol University, Bangkok, NOI
  - King Chulalongkorn Memorial Hospital Chulalongkorn University, Bangkok, Pathumwan
  - Khon Kaen University, Nonthaburi
- United Kingdom (6):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, Edgbaston
  - St Helens & Knowsley Teaching Hospitals, Liverpool, England
  - Chelsea and Westminster Hospital, London, England
  - Newcastle upon Tyne Hospitals, Newcastle upon Tyne, England
  - Manchester University NHSFT, Manchester, London
  - Pinderfields Hospital, Mid Yorkshire NHS Trust, London, West Yorkshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garrel D, Patenaude J, Nedelec B, Samson L, Dorais J, Champoux J, D'Elia M, Bernier J. Decreased mortality and infectious morbidity in adult burn patients given enteral glutamine supplements: a prospective, controlled, randomized clinical trial. Crit Care Med. 2003 Oct;31(10):2444-9. doi: 10.1097/01.CCM.0000084848.63691.1E. PMID 14530749
- [Background] Zhou YP, Jiang ZM, Sun YH, Wang XR, Ma EL, Wilmore D. The effect of supplemental enteral glutamine on plasma levels, gut function, and outcome in severe burns: a randomized, double-blind, controlled clinical trial. JPEN J Parenter Enteral Nutr. 2003 Jul-Aug;27(4):241-5. doi: 10.1177/0148607103027004241. PMID 12903886
- [Background] Peng X, Yan H, You Z, Wang P, Wang S. Effects of enteral supplementation with glutamine granules on intestinal mucosal barrier function in severe burned patients. Burns. 2004 Mar;30(2):135-9. doi: 10.1016/j.burns.2003.09.032. PMID 15019120
- [Derived] Heyland DK, Wibbenmeyer L, Pollack J, Friedman B, Turgeon AF, Eshraghi N, Jeschke MG, Belisle S, Grau D, Mandell S, Velamuri SR, Hundeshagen G, Moiemen N, Shokrollahi K, Foster K, Huss F, Collins D, Savetamal A, Gurney JM, Depetris N, Stoppe C, Ortiz-Reyes L, Garrel D, Day AG; RE-ENERGIZE Trial Team. A Randomized Trial of Enteral Glutamine for Treatment of Burn Injuries. N Engl J Med. 2022 Sep 15;387(11):1001-1010. doi: 10.1056/NEJMoa2203364. Epub 2022 Sep 9. PMID 36082909
- [Derived] Heyland DK, Wischmeyer P, Jeschke MG, Wibbenmeyer L, Turgeon AF, Stelfox HT, Day AG, Garrel D. A RandomizEd trial of ENtERal Glutamine to minimIZE thermal injury (The RE-ENERGIZE Trial): a clinical trial protocol. Scars Burn Heal. 2017 Dec 12;3:2059513117745241. doi: 10.1177/2059513117745241. eCollection 2017 Jan-Dec. PMID 29799545
- See also: Related Info — http://www.criticalcarenutrition.com

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT00985205/SAP_000.pdf